CLINICAL TRIAL: NCT03802734
Title: Perinatal Effects of Mindfulness Phone App Use in Pregnancy (PaMPPr Study)
Acronym: PaMPPr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-048
Record Dates: First submitted 2018-12-20; First posted 2019-01-14 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Sleep; Pregnancy

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Meditation App (Experimental): Group A will be given a free subscription to a mindful meditation phone app for six months. They will also be given an actigraph and a general pregnancy and sleep information leaflet.
  Interventions: Device: Mindful meditation phone app
- No Meditation App (No Intervention): Group B will be given an actigraph and a general pregnancy and sleep information leaflet only.

INTERVENTIONS:
Device: Mindful meditation phone app — Participants in the intervention group will be given a free 6-month subscription to a mindful meditation phone app (Headspace). They will also be given an actigraph and a general pregnancy and sleep information leaflet.
  Arms: Mindful Meditation App

SUMMARY:
There is evidence to show that mindful meditation has a positive impact on health. To date, all the studies done to investigate the effect of mindfulness on pregnancy outcomes have been done through a traditional 8-10 weeks mindfulness classroom program with some home practice. This time-intensive classroom training may be expensive and not convenient for many busy pregnant women. This study will investigate the use of a smartphone app-based intervention to determine if it has the potential to make mindfulness training more accessible, acceptable, and convenient to a larger number of pregnant women. The use of an app as opposed to traditional structured classes may increase a woman's ability and willingness to practice mindfulness because the app can be used almost anywhere and at any time. This pilot study aims to explore the feasibility and acceptability of a smartphone mindfulness meditation application for pregnant women. As well, this study will compare the pregnancy outcomes of women who use the app to those women who do not use the app.

DETAILED DESCRIPTION:
This is a randomised controlled trial to study the effect of the use of a mindfulness meditation app on pregnancy outcomes. This study will measure how often the app is used, as well as indicators of maternal health such as sleep, stress, depression, anxiety and other perinatal outcomes (premature delivery, diabetes during pregnancy (gestational diabetes), high blood pressure in pregnancy (hypertensive disorders of pregnancy), inadequate growth of the baby inside the womb (fetal growth restriction), bleeding in later pregnancy, mode of delivery, pain relief during delivery, length of stay for mother and baby in the hospital, admission of baby in ICU, pain relief medication requirement after delivery, and breastfeeding).

Participants will be randomly assigned to either group A (the experimental group) or group B (the control group). All participants will be given a an actigraph to measure sleep.

Participants in Group A will be given a free subscription to a mindfulness meditation app for six months. They will also be given a general pregnancy sleep leaflet. Participants assigned to Group B will be given the general pregnancy sleep leaflet only.

There will be 3 visits associated with this study. At each of the 3 visits, participants will be given four questionnaires to complete - the Pittsburgh Sleep Quality Index, Perceived Stress Questionnaire, Beck's Anxiety Inventory, and the Edinburgh Postnatal Depression Scale. Participants in Group A will also be asked to complete a fifth survey at their post-partum visit. This survey will collect information on how easy it was to use the mindfulness meditation app.

Information on delivery outcomes will also be collected. This information will include things such as any complications that occur during delivery, baby's birth weight and Apgar score, any complications with baby's health, method of delivery, and pain medications used during delivery.

ELIGIBILITY:
Inclusion Criteria:

* Are able to understand and sign this consent form
* Have a singleton pregnancy (not having twins)
* Are planning to give birth at St. Michael's Hospital
* Have access to personal email, a smartphone, and have a data plan
* Are able to understand and write English
* Are 20-30 weeks into your pregnancy

Exclusion Criteria:

* Are formally practicing a body-mind activity (except yoga) or currently using a mindfulness/meditation app
* Have a known psychiatric diagnosis or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.)
* Have a mood disorder and/or suicide risk
* Have any medical, infectious, or degenerative disease that may affect mood, behavior, and stress levels
* Have a known fetal anomaly
* Have an uncontrolled medical condition that may interfere with sleep or requires immediate treatment
* Have a comorbid sleep disorder, including obstructive sleep apnea, restless legs syndrome, or circadian rhythm sleep disorders
* Are using hypnotic or sedating medications, antidepressant or antipsychotic medications, or currently under psychopharmacological, behavioral, or psychoanalytic treatment
* Are a night shift worker

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 128 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
Sleep | 20 weeks gestation to 6 weeks post partum
  Sleep/wake cycles as measured by an accelerometer that measures tri-axial movement (i.e., actigraphy) for qualitative assessment of sleep.
Use of Meditation Phone App - minutes per day | 20 weeks gestation to 6 weeks post partum
  Measured use of the Headspace app in minutes per day
Use of Meditation Phone App - sessions completed | 20 weeks gestation to 6 weeks post partum
  Measured use of the Headspace app in total number of sessions completed
Use of Meditation Phone App - type of sessions | 20 weeks gestation to 6 weeks post partum
  Breakdown of the number of different session-types used
Use of Meditation Phone App - average session length | 20 weeks gestation to 6 weeks post partum
  Average session length (in minutes)
Use of Meditation Phone App - total time spent meditating | 20 weeks gestation to 6 weeks post partum
  Total number of minutes spent meditating using the meditation phone app

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | PSQI will be completed at 3 time-points: <= 20 weeks gestation, 35-40 weeks gestation, 6 weeks post-partum.
  Participants will rate the frequency of sleep disturbances on a 4-point Likert scale (0 = "Not during the past month"; 1 = "Less than once a week"; 2 = "Once or twice a week"; 3 = "Three or more times a week". Scores will be tallied. A score of 5 or more indicates poor sleep quality. Scores will be compared across 3 time-points.
Perceived Stress Scale (PSS) | PSS will be completed at 3 time-points: <= 20 weeks gestation, 35-40 weeks gestation, 6 weeks post-partum.
  Participants will rate the frequency of certain thoughts and feelings over the past month on a 5-point Likert scale (0 = "Never"; 1 = "Almost never"; 2: "Sometimes"; 3: "Fairly often"; 4: "Very often". Scores will be tallied using the special PSS scoring system. Scores will be compared across 3 time-points.
Edinburgh Postnatal Depression Scale (EPDS) | EDPS will be completed at 3 time-points: <= 20 weeks gestation, 35-40 weeks gestation, 6 weeks post-partum.
  This scale measures post-natal and prenatal depression by asking participants to rate how they have felt emotionally during the last 7 days. Various 4-point Likert scales are used to measure the frequency of occurance (e.g. 0 = No never, 1 = Not very often, 2 = Yes, some of the time, 3 = Yes, most of the time). Scores will be tallied to measure level of depression. Higher scores indicate higher levels of post-natal depression. Scores will be compared across 3 time-points.
Beck Anxiety Inventory (BAI) | 20 weeks gestation to 6 weeks post partum
  Participants will indicate the frequency of anxiety symptoms during the past month on a 4-point Likert scale (0 = No not at all, 1 = Mildly, but it didn't bother me much, 2 = Moderately, it wasn't pleasant at times, 3 = Severely, it bothered me a lot). Scores will be tallied to indicate severity of anxiety. Higher scores indicate higher levels of anxiety. Scores will be compared across 3 time-points.
Complications during pregnancy | Beginning of pregnancy to delivery
  Complications during pregnancy will be recorded using information collected directly from the participant and information collected from their medical chart.
Complications during delivery | Delivery
  Complications during delivery will be recorded using information collected from the patient's medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada